CLINICAL TRIAL: NCT04152083
Title: A Parallel Group, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Eptinezumab Administered Intravenously in Subjects Experiencing an Acute Attack of Migraine
Brief Title: A Study to Evaluate the Efficacy and Safety of Eptinezumab Administered Intravenously in Participants Experiencing Acute Attack of Migraine
Acronym: RELIEF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Collaborators: Alder Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALD403-CLIN-015; 18903A (Other: H. Lundbeck A/S)
Record Dates: First submitted 2019-11-02; First posted 2019-11-05 (Actual); Results first posted 2021-08-16 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — eptinezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eptinezumab (Experimental): Participants will receive a single dose of eptinezumab 100 milligrams (mg) administered via intravenous (IV) infusion on Day 0.
  Interventions: Drug: Eptinezumab
- Placebo (Placebo Comparator): Participants will receive a single dose of placebo matching to eptinezumab administered via IV infusion on Day 0.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eptinezumab — Injection for IV administration
  Arms: Eptinezumab
Drug: Placebo — Injection for IV administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of eptinezumab administered intravenously in participants experiencing an acute attack of migraine.

DETAILED DESCRIPTION:
This will be a parallel group, double-blind, randomized, placebo-controlled study assessing the efficacy of eptinezumab for acute migraine, defined as an active intercurrent migraine occurring in those participants who are candidates for preventive therapy. Participants will be randomized to receive a single dose of eptinezumab or placebo in a 1:1 ratio. The total study duration will be approximately 4 to 12 weeks, including up to an 8-week screening period and 4-week of safety follow-up, with clinic visits occurring on Screening, Day 0 (dosing day), and Week 4.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 1-year history of migraine, with or without aura, with onset of first migraine before age 50.
* Migraine on 4 to 15 days per month in the 3 months prior to screening.
* Headache free for at least 24 hours prior to onset of a qualifying migraine.

Exclusion Criteria:

* Unable to differentiate migraine from other headache or pain disorders.
* Use of the following medication, for any indication, within the 24-hour period prior to dosing with study drug:

  1. triptans, ergotamines and ergot-derivatives
  2. analgesics (including but not limited to acetaminophen, tramadol, nonsteroidal anti-inflammatory drugs [NSAIDs], combination analgesics, caffeine-containing analgesics, and opioids/narcotics) and other acute migraine medication(s)
  3. antiemetic medications (including but not limited to prochlorperazine, promethazine, droperidol, chlorpromazine, metoclopramide)
  4. antihistamines
  5. devices, neuromodulation, neurostimulation, or injectable therapy (trigger point injections, extracranial nerve blocks, facet joint injections, spinal manipulation)
* Use of the following medication, for any indication, in each of the 3 months prior to screening:

  1. opioids/narcotics or butalbital containing products (including combinations) on more than 4 days per month;
  2. triptans, ergotamines, or combination analgesics for 10 or more days per month;
  3. acetaminophen, aspirin or NSAIDs for 15 or more days per month (except if participant is taking 81 mg dose of aspirin for cardiac prophylaxis)
* History or diagnosis of chronic tension-type headache, hypnic headache, cluster headache, hemicrania continua, new daily persistent headache, or unusual migraine subtypes such as hemiplegic migraine (sporadic and familial), ophthalmoplegic migraine and migraine with neurological accompaniments that are not typical of migraine aura (for example, diplopia, altered consciousness, or long duration).
* Any changes to preventive migraine treatment(s) within 1 month prior to screening and up to treatment with the study drug (Day 0).
* Any use of approved devices, neuromodulation, neurostimulation, or injectable therapy (trigger point injections, extracranial nerve blocks, facet joint injections) within the 24-hour period prior to treatment with study drug (Day 0).
* Any use of botulinum toxin for migraine or for any other medical/cosmetic reasons requiring injections within 7 days prior to treatment with study drug (Day 0).
* Any use of systemic corticosteroid for migraine or any other reason within 3 months prior to treatment with study drug (Day 0).
* Evidence or medical history of clinically significant psychiatric diseases that are uncontrolled and/or untreated.
* Receipt of any monoclonal antibody treatment, for migraine or any other indication, (within or outside a clinical study) within 6 months prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (57):
- United States (52):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Advanced Research Center, Anaheim, California
  - The Neurology Center of Southern California - Carlsbad, Carlsbad, California
  - Excell research Inc, Oceanside, California
  - Anderson Clinical Research, Redlands, California
  - University of Colorado Hospital, Aurora, Colorado
  - Denver Neurological Clinic - Denver, Denver, Colorado
  - Coastal Connecticut Research LLC, New London, Connecticut
  - Ki Health Partners LLC, dba New England Institute for Clinical Research, Stamford, Connecticut
  - The George Washington Medical Faculty Associates, Washington D.C., District of Columbia
  - Medicinae Doctor Clinical, Hallandale, Florida
  - AGA Clinical trials, Hialeah, Florida
  - Meridien Research - Maitland, Maitland, Florida
  - Palm Beach Neurology and Premiere Research Institute, West Palm Beach, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Office of Doctor Frank Berenson, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Meridian Clinical Research - Savannah Neurology Specialists, Savannah, Georgia
  - Cedar Crosse Research Center, Chicago, Illinois
  - College Park Family Care Center Physicians, Overland Park, Kansas
  - Phoenix Medical Research, Prairie Village, Kansas
  - Central Kentucky Research Associates, Lexington, Kentucky
  - Boston Clinical Trials, Boston, Massachusetts
  - MedVadis Research Corporation, LLC, Waltham, Massachusetts
  - Michigan Head Pain and Neurological institute, Ann Arbor, Michigan
  - Clinical Research Institute - Minneapolis, Minneapolis, Minnesota
  - Headache Neurology Research Institute, Ridgeland, Mississippi
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinvest Research, Springfield, Missouri
  - Nevada Headache Institute, Las Vegas, Nevada
  - Albuqerque Clinical Trials, Albuquerque, New Mexico
  - Dent Neurologic Institute - Amherst, Amherst, New York
  - Integrative Clinical Trials, Brooklyn, New York
  - CTI Clinical Research center, Cincinnati, Ohio
  - Aventiv Research - Columbus, Columbus, Ohio
  - Hometown Urgent Care And Research - Huber Heights, Dayton, Ohio
  - Neuro-Behavioral Clinical Research Inc, North Canton, Ohio
  - Delricht Research, Tulsa, Oklahoma
  - Summit Research Network, Portland, Oregon
  - Frontier Clinical Rsearch LLC, Smithfield, Pennsylvania
  - Coastal Carolina Research Center - Mount Pleasant, Mt. Pleasant, South Carolina
  - Chattanooga Medical research LLC, Chattanooga, Tennessee
  - WR-ClinSearch LLC, Chattanooga, Tennessee
  - Holston Medical Group - Kingsport, Kingsport, Tennessee
  - Ventavia Research Group, LLC, Fort Worth, Texas
  - Texas Center for Drug Development Inc, Houston, Texas
  - Ventavia Research Group, LLC, Keller, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
  - Neuroscience Group, Neenah, Wisconsin
- Georgia (5):
  - Ltd "Acad Fridon Todua Medical Center - Ltd Research Institute of Clinical Medicine", Tbilisi
  - Ltd "Aversi Clinic", Tbilisi
  - Ltd "Multiprofile Clinica Consilium Medulla", Tbilisi
  - Ltd Simon Khechinashvili University Clinic, Tbilisi
  - td "Israel-Georgia Medical Research Clinic Helsicore", Tbilisi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cady R, Lipton RB, Buse DC, Josiassen MK, Lindsten A, Ettrup A. Optimization of acute medication use following eptinezumab initiation during a migraine attack: post hoc analysis of the RELIEF study. J Headache Pain. 2022 Jul 28;23(1):91. doi: 10.1186/s10194-022-01463-3. PMID 35902796
- [Derived] Ailani J, McAllister P, Winner PK, Chakhava G, Krog Josiassen M, Lindsten A, Sperling B, Ettrup A, Cady R. Rapid resolution of migraine symptoms after initiating the preventive treatment eptinezumab during a migraine attack: results from the randomized RELIEF trial. BMC Neurol. 2022 Jun 3;22(1):205. doi: 10.1186/s12883-022-02714-1. PMID 35659622
- [Derived] McAllister P, Winner PK, Ailani J, Buse DC, Lipton RB, Chakhava G, Josiassen MK, Lindsten A, Mehta L, Ettrup A, Cady R. Eptinezumab treatment initiated during a migraine attack is associated with meaningful improvement in patient-reported outcome measures: secondary results from the randomized controlled RELIEF study. J Headache Pain. 2022 Feb 7;23(1):22. doi: 10.1186/s10194-021-01376-7. PMID 35130832
- [Derived] Winner PK, McAllister P, Chakhava G, Ailani J, Ettrup A, Krog Josiassen M, Lindsten A, Mehta L, Cady R. Effects of Intravenous Eptinezumab vs Placebo on Headache Pain and Most Bothersome Symptom When Initiated During a Migraine Attack: A Randomized Clinical Trial. JAMA. 2021 Jun 15;325(23):2348-2356. doi: 10.1001/jama.2021.7665. PMID 34128999

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to receive either 100 milligrams (mg) eptinezumab or placebo in a 1:1 ratio.
Groups:
- Eptinezumab: Participants received a single dose of eptinezumab 100 mg administered via intravenous (IV) infusion on Day 0.
- Placebo: Participants received a single dose of placebo matched to eptinezumab administered via IV infusion on Day 0.
Period: Overall Study
Arm/Group | Eptinezumab | Placebo
Started | 241 | 244
Received at Least 1 Dose of Study Drug | 238 | 242
Completed | 235 | 241
Not Completed | 6 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Randomized but not treated | 3 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received eptinezumab or placebo.
Groups:
- Eptinezumab: Participants received a single dose of eptinezumab 100 mg administered via IV infusion on Day 0.
- Total: Total of all reporting groups
Arm/Group | Eptinezumab | Placebo | Total
Number analyzed (Participants) | 238 | 242 | 480
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (11.99) | 44.1 (12.12) | 44.5 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202 | 201 | 403
  Male | 36 | 41 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 31 | 60
  Not Hispanic or Latino | 209 | 211 | 420
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 200 | 213 | 413
  Race: Black or African American | 30 | 19 | 49
  Race: Asian | 2 | 3 | 5
  Race: American Indian or Alaska Native | 2 | 1 | 3
  Race: Native Hawaiian or other Pacific Islander | 1 | 1 | 2
  Race: Other | 0 | 1 | 1
  Race: Multiple | 3 | 4 | 7
Number of Migraine Days/Month [Mean (Standard Deviation); unit: days/month] — Average number of migraine days per month during the 3 months prior to screening is reported. Each month consisted of 28 days.
  days/month | 7.2 (2.65) | 7.2 (2.56) | 7.2 (2.60)
Number of Participants With Most Bothersome Symptoms (MBS) [Number; unit: participants]
  Photophobia | 114 | 114 | 228
  Nausea | 78 | 79 | 157
  Phonophobia | 46 | 47 | 93
  Missing | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to Headache Pain Freedom
Description: Time to headache pain freedom defined as the time that the participant reported freedom of pain, meaning their headache pain had gone from moderate to severe at baseline to no pain.
Time Frame: Up to 48 hours postdose
Population: Full analysis population (FAP) included all randomized participants who received eptinezumab or placebo.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 238 | 242
hours | 4.0 [2.5 to 12.0] | 9.0 [3.0 to 48.0]
Statistical Analysis 1: Comparison: Eptinezumab vs Placebo; The median estimate for each treatment group, hazard ratio, and its 95% confidence interval (CI) were based on the stratified Cox model with Efron's method of tie handling. The analysis was censored at the time point of first rescue medication. The stratification factors were concomitant migraine preventive treatment use and region; Test type: Other; p = 0.0006, Likelihood ratio test — Threshold for significance at 0.05 level; Hazard Ratio (HR) = 1.54, 95% CI 2-sided [1.20 to 1.98]

2. Primary Outcome: Time to Absence of Most Bothersome Symptom (MBS)
Description: Time to absence of most bothersome symptom defined as the time that the participant reported absence of MBS (of nausea, photophobia, or phonophobia).
Time Frame: Up to 48 hours postdose
Population: FAP included all randomized participants who received eptinezumab or placebo. Here, 'Overall number of participants analyzed' signifies participants with both baseline and post-baseline data (the symptom that was most bothersome).
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 238 | 240
hours | 2.0 [1.0 to 3.5] | 3.0 [1.5 to 12.0]
Statistical Analysis 1: Comparison: Eptinezumab vs Placebo; The median estimate for each treatment group, hazard ratio, and its 95% CI were based on the stratified Cox model with Efron's method of tie handling. The analysis was censored at the time point of first rescue medication. The stratification factors were concomitant migraine preventive treatment use and region; Test type: Other; p < 0.0001, Likelihood ratio test — Threshold for significance at 0.05 level; Hazard Ratio (HR) = 1.75, 95% CI 2-sided [1.41 to 2.19]

3. Secondary Outcome: Headache Pain Freedom at 2 Hours
Description: Number of participants with freedom from headache pain at 2 hours postdose are reported. Freedom from headache pain meaning that the headache pain that had gone from moderate to severe at baseline to no pain with no administration of rescue medications.
Time Frame: 2 hours
Population: FAP included all randomized participants who received eptinezumab or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 238 | 242
Participants | 56 | 29
Statistical Analysis 1: Comparison: Eptinezumab vs Placebo; Odds ratio and 95% CI were based on Cochran-Mantel-Haenszel (CMH) test adjusted for the study's stratification factors of concomitant migraine preventive treatment use and region; Test type: Other; p = 0.0009, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Odds Ratio (OR) = 2.27, 95% CI 2-sided [1.39 to 3.72]

4. Secondary Outcome: Absence of MBS at 2 Hours
Description: Number of participants with absence of MBS (of nausea, photophobia, or phonophobia) at 2 hours postdose are reported.
Time Frame: 2 hours
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 238 | 240
Participants | 132 | 86
Statistical Analysis 1: Comparison: Eptinezumab vs Placebo; Odds ratio and 95% CI were based on CMH test adjusted for the study's stratification factors of concomitant migraine preventive treatment use and region; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Odds Ratio (OR) = 2.25, 95% CI 2-sided [1.55 to 3.25]

5. Secondary Outcome: Headache Pain Freedom at 4 Hours
Description: Number of participants with freedom from headache pain at 4 hours postdose are reported. Freedom from headache pain meaning that the headache pain that had gone from moderate to severe at baseline to no pain with no administration of rescue medications.
Time Frame: 4 hours
Population: FAP included all randomized participants who received eptinezumab or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 238 | 242
Participants | 111 | 64

6. Secondary Outcome: Absence of MBS at 4 Hours
Description: Number of participants with absence of MBS (of nausea, photophobia, or phonophobia) at 4 hours postdose are reported.
Time Frame: 4 hours
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 238 | 240
Participants | 155 | 90

7. Secondary Outcome: Use of Rescue Medication Within the First 24 Hours
Description: Rescue medication was defined as any medication to treat migraine or migraine-associated symptoms, which could have been provided to the participant any time after 2 hours post-start of infusion. Use of rescue medication was captured in the eDiary. Number of participants who used rescue medication up to 24 hours postdose are reported.
Time Frame: Up to 24 hours postdose
Population: FAP included all randomized participants who received eptinezumab or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Eptinezumab | Placebo
Number analyzed (Participants) | 238 | 242
Participants | 75 | 145

ADVERSE EVENTS:
Time Frame: Start of treatment (Day 0) through end of study (Week 4)
Description: Safety population included all participants who received eptinezumab or placebo.
Arm/Group | Eptinezumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/238 | 0/242
Serious Adverse Events (participants affected / at risk) | 0/238 | 0/242
Other Adverse Events (participants affected / at risk) | 5/238 | 0/242
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eptinezumab (N=238) | Placebo (N=242)
Hypersensitivity (Immune system disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT04152083/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT04152083/SAP_001.pdf